CLINICAL TRIAL: NCT04238065
Title: A Phase 3 Randomized, Single-blind, Multicenter, Clinical Control Study to Evaluate the Efficacy and Safety of Caterna Virtual Reality Facilitating Treatment Patients With Amblyopia in Children
Brief Title: A Clinical Trial of Caterna Virtual Reality Facilitating Treatment in Children With Amblyopia
Acronym: VRTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Shijing Medical Software (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Beijing University (Unknown); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GuangzhouShijingMS
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Amblyopia
Keywords: Amblyopia; Virtual Reality
MeSH Terms: conditions — Amblyopia | interventions — Transdermal Patch; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: One arm receive VR treatment while the other arm does not. Both arms get best optical correction and 2 hours (for mild and moderate amblyopia）patch or 6 hours (for severe amblyopia) patch their non-amblyopia eyes.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Research centers are used as a stratification factor. The researchers include subjects in the trial group or control group based on randomized envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR treatment (Experimental): The arm will use the virtual reality headset reproduces dynamic video content with perceptual learning and binocular perception (including stereopsis) that is visually perceived a little bit faster, brighter, and higher contrast to the amblyopia eyes .
  The each VR therapy length is 30 minutes with 5 minute break after 15 minutes' therapy sequence, 3 times per week, total 13 weeks.
  All amblyopia eyes are best optical correction or combining patching non-amblyopia eyes if there're more than 2 lines difference best corrected vision acuity.
  Interventions: Device: Caterna Virtual Reality; Device: Spectacles(Best optical corrected distance vision); Device: Patch
- control (Placebo Comparator): This arm of amblyopia eyes are all best optical correction or combining patching non-amblyopia eyes if there're more than 2 lines difference best corrected vision acuity.
  No VR therapy.
  Interventions: Device: Spectacles(Best optical corrected distance vision); Device: Patch

INTERVENTIONS:
Device: Caterna Virtual Reality — Vivid interactive games of perceptual learning content, with artificial intelligent sound and scores to feedback vision and actions results, which can be connected to the supervision of cellphone software"Wechat" to upload vision acuity and choose 2 eyes' video output automaticly.
  Other Names: SJ-VRS2018; DOBOSO VR; Vision Therapy Software
  Arms: VR treatment
Device: Spectacles(Best optical corrected distance vision) — Each eye has best corrected vision spectacles with best corrected optical lens.
  Other Names: Optical correction
Device: Patch — 2 hours patch to the non-amblyopia eye if the other amblyopia eye is mild or moderate amblyopia; 6 hours patch to the non-amblyopia eye if the other amblyopia eye is severe abmlyopia
  Other Names: Occlusion

SUMMARY:
It aims to find the effectiveness and the safety of Virtual Reality (Caterna, DOBOSO, item code: SJ-VRS2018) to facilitate amblyopia treatment combining spectacles and occlusion. And it also aims to test whether amblyopia treatment outcomes with spectacles, occlusion and VR are significant better than those without VR, but with spectacles and occlusion.

The experiment arm is designed to use the Caterna VR to treat amblyopia for total consistent 13 weeks, 3 times per week, while the control arm is not.

Both arms are best optical correction and with patch the non-amblyopia eye 2 hours or 6 hours per day.

All eyes are followed up for total 13 weeks.

DETAILED DESCRIPTION:
The amblyopia eye will see the video content from Caterna VR a little bit earlier (12 ms) than the other non-amblyopia eye.

Also, the illumination and contrast are both adjusted to balance 2 eyes' clarity.

One VR treatment sequence is 30 minutes with 5 minutes break in the middle.

ELIGIBILITY:
Inclusion Criteria:

1. Ages from 4~12 years old (including 4 years or 12 years old）；
2. According to the Chinese Medical Association Ophthalmology branch: Strabismus and Pediatric Ophthalmology Experts "Consensus of Amblyopia Diagnosis " (2011) as the standard to be diagnosed as amblyopia with abnormal vision than that of age-based norms, that is, caused by abnormal visual development due to strabismus, uncorrected refractive error or form deprivation, the best corrected vision acuity of single eye or both eyes below age-based norms; Or 2 eyes' vision acuity difference larger than 2 lines or more. The normal minimum limit of vision acuity for children of different ages are as the followings: The normal minimum limit of vision acuity for children aged 4 to 5 years is 0.5 (decimal vision acuity); And the normal minimum limit of vision acuity for children aged 6 and over is 0.7(decimal vision acuity).
3. The subject's supervision is fully understand the purpose of the trial and sign an informed consent form; And the subject can cooperate with the whole treatment and related eye examinations。 -

Exclusion Criteria:

1. Subjects suffered from tumors, heart disease, hypertension (blood pressure top limitation of children aged 4 to 6 years: 110/70 mmHg, blood pressure top limitation of children aged 7 to 12 years: 120/80 mmHg), or epilepsy;
2. The subject has implanted electronic devices, such as pacemakers, etc.
3. The subject had or has a mental illness;
4. Any eye of the subject due to keratitis, conjunctivitis, internal turning eyelashes and other diseases leading to photophobia or continuing tears;
5. Subject suffered from vertigo, acrophobia or traumatic brain lesions;
6. The subject's eye has congenital glaucoma, congenital ptosis, dacryocystitis, trauma and other significant vision related lesions;
7. Subject received a masking therapy or a treatment instrument for amblyopia treatment before joining this study;
8. The subject participated in other clinical trials before joining this study;
9. For safety reasons or for the benefit of patients, the researchers believe that the patient should not participate in other conditions, such as suffering from a certain severe heart, liver or kidney disease.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of amblyopia treatment with VR | 13 weeks
  General Effectiveness=Number of both cured eyes and effective eyes from total number×100%

SECONDARY OUTCOMES:
Effectiveness of 8 weeks' VR amblyopia treatment | 8 weeks
  General Effectiveness=Number of both cured eyes and effective eyes from total number×100%
Effectiveness of 4 weeks' VR amblyopia treatment | 4 weeks
  General Effectiveness=Number of both cured eyes and effective eyes from total number×100%
Stereopsis: distance and near, respectively | 13 weeks
  Ratio of stereopsis perception=(Number of stereopsis perception /Total number)*100%
Contrast sensitivity function(CSF) | 13 weeks
  Difference between those final CSF and baseline CSF

OTHER OUTCOMES:
Severe Adverse Event Number | 13 weeks
  Total number of Severe Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Liu, Study Director — Guangzhou Shijing Medical Software; Mosheng Zhou, Study Chair — Guangzhou Shijing Medical Software
Locations (4):
- China (4):
  - the first affiliated hospital of Beijing University, Beijing, Beijing Municipality
  - Guangzhou Shijing Medical Software Co., Ltd., Guangzhou, Guangdong
  - Zhongshan Ophthalmic center, Sun Yat-sen University, Guanzhou, Guangdong
  - The first affiliated hospital of Nanjing University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Repka MX, Beck RW, Holmes JM, Birch EE, Chandler DL, Cotter SA, Hertle RW, Kraker RT, Moke PS, Quinn GE, Scheiman MM; Pediatric Eye Disease Investigator Group. A randomized trial of patching regimens for treatment of moderate amblyopia in children. Arch Ophthalmol. 2003 May;121(5):603-11. doi: 10.1001/archopht.121.5.603. PMID 12742836
- [Result] Holmes JM, Kraker RT, Beck RW, Birch EE, Cotter SA, Everett DF, Hertle RW, Quinn GE, Repka MX, Scheiman MM, Wallace DK; Pediatric Eye Disease Investigator Group. A randomized trial of prescribed patching regimens for treatment of severe amblyopia in children. Ophthalmology. 2003 Nov;110(11):2075-87. doi: 10.1016/j.ophtha.2003.08.001. PMID 14597512
- [Result] Scheiman MM, Hertle RW, Beck RW, Edwards AR, Birch E, Cotter SA, Crouch ER Jr, Cruz OA, Davitt BV, Donahue S, Holmes JM, Lyon DW, Repka MX, Sala NA, Silbert DI, Suh DW, Tamkins SM; Pediatric Eye Disease Investigator Group. Randomized trial of treatment of amblyopia in children aged 7 to 17 years. Arch Ophthalmol. 2005 Apr;123(4):437-47. doi: 10.1001/archopht.123.4.437. PMID 15824215
- [Result] Yazdani N, Sadeghi R, Momeni-Moghaddam H, Zarifmahmoudi L, Ehsaei A, Barrett BT. Part-time versus full-time occlusion therapy for treatment of amblyopia: A meta-analysis. J Curr Ophthalmol. 2017 Mar 6;29(2):76-84. doi: 10.1016/j.joco.2017.01.006. eCollection 2017 Jun. PMID 28626815
- [Result] Jin H, Yi JL, Xie H, Xiao F, Wang WJ, Shu XM, Xu YL, Chen SL, Ye WX. [A study on visual development among preschool children]. Zhonghua Yan Ke Za Zhi. 2011 Dec;47(12):1102-6. Chinese. PMID 22336120
- [Result] He MG. [The quality of epidemiological research on pediatric refractive error and amblyopia in China needs to be improved]. Zhonghua Yan Ke Za Zhi. 2017 Jan 11;53(1):3-6. doi: 10.3760/cma.j.issn.0412-4081.2017.01.002. Chinese. PMID 28162193